CLINICAL TRIAL: NCT05768828
Title: Calcitonin Gene-Related Peptide (CGRP) and Neurophysiological Biomarkers of Migraine
Brief Title: Stimulation-evoked Calcitonin Gene-Related Peptide (CGRP) as Biomarker of Migraine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: BB 040/22
Record Dates: First submitted 2023-03-03; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood from cubital vein and lacrimal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Migraine: Patients suffering from migraine based on ICHD-3 criteria
  Interventions: Diagnostic Test: Nociceptive Blink Reflex
- Controls: Patients free of headaches or not suffering from headaches with a frequency that exceeds 1x/year
  Interventions: Diagnostic Test: Nociceptive Blink Reflex

INTERVENTIONS:
Diagnostic Test: Nociceptive Blink Reflex — Noxious trigeminal electrical stimulation at different interstimulus intervals using 1.5x the pain threshold in order to provoke a release of trigeminal CGRP

SUMMARY:
This study aims to improve the management migraine by providing a more profound understanding of the interactions of pain disinhibition on the brain stem level and calcitonin gene-related peptide as a main mediator in the generation of migraine headaches. For this purpose, this observational study investigates established neurophysiological and blood biomarkers parameters in association with the clinical phenotype.

DETAILED DESCRIPTION:
The study's focus is the investigation of mechanisms that are directly related to the pain generation in migraine. In this context, the primary endpoint is an enhancement of trigeminal stimulation evoked calcitonin gene-related peptide (CGRP). The stimulation is normalized using an established protocol to elicit the nociceptive blink reflex, which is a brain stem reflex to study the trigemino-spinal system. We expect CGRP levels to rise more in patients affected by migraine as compared to controls, based on the observation that painful stimulation elicits migraine attacks. Furthermore, baseline CGRP levels and their association with markers of brainstem excitability are probed.

ELIGIBILITY:
Inclusion Criteria:

* Migraine according to ICHD-3 criteria (cases)
* No headaches or tension-type headache frequency <1x/year (controls)

Exclusion Criteria:

* other chronic pain disorder

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited through the outpatient headache department and through public adverstisement. Patients are consecutively recruited and inclusion/exclusion criteria are minimzied to avoid selection bias.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Plasma levels of Calcitonin Gene-Related Peptide | cross-sectional, once after stimulation
  Plasma levels of Calcitonin Gene-Related Peptide from samples taken from the cubital vein following nociceptive trigeminal stimulation

SECONDARY OUTCOMES:
Lacrimal fluid levels of Calcitonin Gene-Related Peptide | cross-sectional, once after stimulation
  Lacrimal fluid levels of Calcitonin Gene-Related Peptide from samples taken from the outer angle of the eye following nociceptive trigeminal stimulation
Habituation of the nociceptive blink reflex in correlation with plasma levels of Calcitonin Gene-Related Peptide | cross-sectional, once before stimulation
  Explore the correlation of the amplitude of the R2 component of the nociceptive blink reflex with baseline plasma levels of Calcitonin Gene-Related Peptide
Habituation of the nociceptive blink reflex in correlation with lacrimal fluid levels of Calcitonin Gene-Related Peptide | cross-sectional, once before stimulation
  Explore the correlation of the amplitude of the R2 component of the nociceptive blink reflex with baseline lacrimal fluid levels of Calcitonin Gene-Related Peptide

CONTACTS AND LOCATIONS:
Locations (1):
- University Medicine Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No
IPD can be shared upon reasonable request. Data protection regulation preclude public sharing of data.